CLINICAL TRIAL: NCT02236988
Title: A Phase 1, Open-Label, Single Center Study to Evaluate the Pharmacokinetics of Prototype Modified-Release Formulations Of Apremilast (CC-10004) in Healthy Male Subjects
Brief Title: Study to Evaluate Pharmacokinetics of Prototype Modified-Release Formulations Of Apremilast in Healthy Men
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CC-10004-CP-027
Expanded Access: NCT03740516 (No longer available)
Record Dates: First submitted 2014-09-09; First posted 2014-09-11 (Estimated); Results first posted 2021-06-01 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-03

CONDITIONS: Healthy Volunteers
Keywords: Apremilast; Healthy male subjects; Pharmacokinetics
MeSH Terms: interventions — apremilast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1 (Experimental): Participants received the following 4 treatments, given in 4 possible sequences (ADBC, BACD, CBDA, and DCAB) with 7 to 10 days between each treatment:
  A) Two oral doses of 30 mg apremilast immediate release tablets 12 hours apart (reference formulation) B) A single oral dose 75 mg apremilast tablet prototype MR 1 C) A single oral dose 75 mg apremilast tablet prototype MR 2 D) A single oral dose 75 mg apremilast capsule prototype MR 3
  Interventions: Drug: Apremilast Immediate Release; Drug: Apremilast Modified Release 1; Drug: Apremilast Modified Release 2; Drug: Apremilast Modified Release 3
- Group 2 (Experimental): Participants received the following 4 treatments, given in 4 possible sequences (AGEF, EAFG, FEGA, and GFAE) with 7 to 10 days between each treatment:
  A) Two oral doses of 30 mg apremilast immediate release tablets 12 hours apart (reference formulation) E) A single oral dose 75 mg apremilast capsule prototype MR 4 F) A single oral dose 75 mg apremilast capsule prototype MR 5 G) A single oral dose 75 mg apremilast capsule prototype MR 6
  Interventions: Drug: Apremilast Immediate Release; Drug: Apremilast Modified Release 4; Drug: Apremilast Modified Release 5; Drug: Apremilast Modified Release 6
- Group 3 (Experimental): Participants received the following 3 treatments, given in 6 possible sequences (AIJ, IJA, JAI, AJI, IAJ, or JIA) with 7 to 10 days between each treatment:
  A) Two oral doses of 30 mg apremilast immediate release tablets 12 hours apart (reference formulation) I) A single oral dose 80 mg apremilast capsule prototype MR 8 J) A single oral dose 80 mg apremilast capsule prototype MR 9
  Interventions: Drug: Apremilast Immediate Release; Drug: Apremilast Modified Release 8; Drug: Apremilast Modified Release 9
- Group 4 (Experimental): Participants received the following 5 treatments, given in 10 possible sequences (ALOMN, LMANO, MNLOA, NOMAL, OANLM, NMOLA, ONAML, AOLNM, LAMON, or MLNAO) with 7 to 10 days between each treatment:
  A) Two oral doses of 30 mg apremilast immediate release tablets 12 hours apart (reference formulation) L) A single oral dose 80 mg apremilast capsule prototype MR 11 M) A single oral dose 80 mg apremilast capsule prototype MR 12 N) A single oral dose 80 mg apremilast capsule prototype MR 13 O) A single oral dose 80 mg apremilast capsule prototype MR 14
  Interventions: Drug: Apremilast Immediate Release; Drug: Apremilast Modified Release 11; Drug: Apremilast Modified Release 12; Drug: Apremilast Modified Release 13; Drug: Apremilast Modified Release 14

INTERVENTIONS:
Drug: Apremilast Immediate Release — 30 mg immediate release tablets
  Other Names: Otezla; CC-10004
Drug: Apremilast Modified Release 1 — 75 mg oral tablet of prototype modified release (MR) 1
  Arms: Group 1
Drug: Apremilast Modified Release 2 — 75 mg oral tablet of prototype MR 2
  Arms: Group 1
Drug: Apremilast Modified Release 3 — 75 mg oral capsule of prototype MR 3
  Arms: Group 1
Drug: Apremilast Modified Release 4 — 75 mg oral capsule of prototype MR 4
  Arms: Group 2
Drug: Apremilast Modified Release 5 — 75 mg oral capsule of prototype MR 5
  Arms: Group 2
Drug: Apremilast Modified Release 6 — 75 mg oral capsule of prototype MR 6
  Arms: Group 2
Drug: Apremilast Modified Release 8 — 80 mg oral capsule of prototype MR 8
  Arms: Group 3
Drug: Apremilast Modified Release 9 — 80 mg oral capsule of prototype MR 9
  Arms: Group 3
Drug: Apremilast Modified Release 11 — 80 mg oral capsule of prototype MR 11
  Arms: Group 4
Drug: Apremilast Modified Release 12 — 80 mg oral capsule of prototype MR 12
  Arms: Group 4
Drug: Apremilast Modified Release 13 — 80 mg oral capsule of prototype MR 13
  Arms: Group 4
Drug: Apremilast Modified Release 14 — 80 mg oral capsule of prototype MR 14
  Arms: Group 4

SUMMARY:
This study will assess up to 12 different oral formulations of apremilast to determine how much apremilast is absorbed by the body compared to a reference formulation.

DETAILED DESCRIPTION:
This will be a single-center, open-label, crossover, single modified-release-dose study in adult males to evaluate the pharmacokinetics (PK) of prototype modified-release (MR) formulations compared to the reference immediate-release (IR) apremilast formulation. Within 4 separate groups, participants will be randomly assigned to a treatment sequence. A total of up to 12 test MR formulations may be evaluated.

Group 1: A 4-sequence, 4-period design to compare three modified-release prototypes with the reference immediate-release formulation. A total of 16 participants will be enrolled to obtain at least 12 participants who complete all 4 periods.

Group 2: A 4-sequence, 4-period design to compare three MR prototypes with the reference IR formulation. Sixteen participants will be enrolled to obtain at least 12 participants who complete all four periods.

Group 3: A six-sequence, three-period design to compare two MR prototypes with the reference IR formulation. Eighteen participants will be enrolled to obtain at least 12 participants who complete all three periods.

Group 4: A 10-sequence, 5-period design to compare four MR prototypes with the reference IR formulation. Thirty participants will be enrolled to obtain at least 20 participants who complete all five periods.

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy ALL of the following criteria to be eligible for enrollment into the study:

1. Must understand and voluntarily sign a written informed consent form prior to any study-related procedures being performed.
2. Must be able to communicate with the investigator, understand and comply with the requirements of the study, and agree to adhere to restrictions and examination schedules.
3. Male subjects of any race between 18 to 55 years of age (inclusive), and in good health as determined by the Investigator.
4. Has a body mass index between 18 and 33 kg/m^2 (inclusive).
5. No clinically significant laboratory tests as determined by the investigator.
6. Must not have a fever, with systolic blood pressure: 90 to 140 mmHg and diastolic blood pressure: 60 to 90 mmHg, and pulse rate: 40 to 110 bpm (measurements taken while lying down).
7. Must have a normal or clinically acceptable 12-lead electrocardiogram (ECG).
8. Subjects (including those who have had a vasectomy) who engage in activity in which conception is possible must use barrier contraception (male latex condom or non-latex condom not made out of natural [animal] membrane [eg, polyurethane]) while on study medication, and for 28 days after the last dose of study medication.
9. Must agree to refrain from donating sperm, blood or plasma (other than for this study) while participating in this study and for at least 28 days after the last dose of study drug.

Exclusion Criteria:

The presence of ANY of the following will exclude any healthy subject from enrollment into the study:

1. History of any clinically significant and relevant neurological, gastrointestinal, renal, hepatic, cardiovascular, psychological, pulmonary, metabolic, endocrine, hematological, allergic disease, drug allergies, or other major disorders.
2. Any condition which places the subject at unacceptable risk if he were to participate in the study, or confounds the ability to interpret data from the study.
3. Use of any prescribed systemic or topical medication within 30 days of the first dose administration, unless Sponsor agreement is obtained.
4. Use of any non-prescribed systemic or topical medication (including vitamin/mineral supplements, and herbal medicines) within 14 days of the first dose administration, unless Sponsor agreement is obtained.
5. Any surgical or medical condition possibly affecting drug absorption, distribution, metabolism and excretion, eg, bariatric procedure, colon resection, irritable bowel syndrome, Crohn's disease, etc. Subjects with cholecytectomy and appendectomy may be included.
6. Exposure to an investigational drug (new chemical entity) within 30 days prior to the first dose administration or 5 half-lives of that investigational drug, if known (whichever is longer).
7. Donated blood or plasma within 8 weeks before the first dose administration to a blood bank or blood donation center.
8. History of drug abuse (as defined by the current version of the Diagnostic and Statistical Manual (DSM) within 2 years before dosing, or a positive drug screen reflecting consumption of illicit drugs.
9. History of alcohol abuse (as defined by the current version of the DSM) within 2 years before dosing, or a positive alcohol screen.
10. Known to have serum hepatitis, or known to be a carrier of the hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV) antibody, or have a positive result to the test for human immunodeficiency virus (HIV) antibodies at Screening.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2014-01-07 (Actual); Primary Completion 2014-09-11 (Actual); Study Completion 2014-09-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (1):
- Covance Clinical Research Unit Inc., Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at a single study site in the United States from July 2013 to September 2014.
Pre-assignment Details: This was an open-label crossover study that consisted of 4 groups of participants and tested 12 different modified release (MR) formulations of apremilast versus the reference immediate release (IR) formulation. Within each group participants were randomized to a treatment sequence.
Period: Overall Study
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Started | 16 | 16 | 18 | 30
Completed | 16 | 16 | 18 | 27
Not Completed | 0 | 0 | 0 | 3
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Unable to Comply with Study Visits | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Total
Number analyzed (Participants) | 16 | 16 | 18 | 30 | 80
Age, Continuous [Mean (Full Range); unit: years] | 39.1 [29 to 55] | 34.1 [20 to 50] | 30.4 [21 to 43] | 33.3 [20 to 55] | 34.0 [20 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 16 | 16 | 18 | 30 | 80
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 3 | 2 | 7
  Not Hispanic or Latino | 16 | 14 | 15 | 28 | 73
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 11 | 12 | 16 | 21 | 60
  Black or African American | 3 | 3 | 2 | 5 | 13
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1
  Asian | 1 | 1 | 0 | 3 | 5
  Other | 0 | 0 | 0 | 1 | 1
Body Mass Index (BMI) [Mean (Full Range); unit: kg/m^2] | 26.82 [22.5 to 31.6] | 25.56 [21.7 to 29.1] | 24.83 [20.2 to 31.2] | 25.15 [20.3 to 32.4] | 25.49 [20.2 to 32.4]

OUTCOME MEASURES:

1. Primary Outcome: Group 1: Observed Maximum Plasma Concentration (Cmax) of Apremilast
Description: Concentrations of apremilast in plasma were measured using a validated liquid chromatography tandem mass spectrometry assay.
Time Frame: IR reference formulation: predose and at 0.5, 1, 2, 3, 5, 8, 12, 12.5, 13, 14, 15, 17, 20, 24, 36, 48, 60, and 72 hours after the first dose; MR formulations: predose and at 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 14, 16, 20, 24, 30, 36, 48, and 72 hours postdose.
Population: The pharmacokinetic (PK) population included all participants who received at least one dose of apremilast and had evaluable PK profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Group 1: Apremilast Immediate Release: Participants received two oral doses of 30 mg apremilast immediate release tablets 12 hours apart (reference formulation).
- Group 1: Apremilast Modified Release 1: Participants received a single oral dose 75 mg apremilast tablet prototype MR 1.
- Group 1: Apremilast Modified Release 2: Participants received a single oral dose 75 mg apremilast tablet prototype MR 2.
- Group 1: Apremilast Modified Release 3: Participants received a single oral dose 75 mg apremilast capsule prototype MR 3.
Arm/Group | Group 1: Apremilast Immediate Release | Group 1: Apremilast Modified Release 1 | Group 1: Apremilast Modified Release 2 | Group 1: Apremilast Modified Release 3
Number analyzed (Participants) | 16 | 16 | 16 | 16
ng/mL | 409.96 (34.9) | 267.85 (56.4) | 329.78 (52.2) | 345.11 (41.5)
Statistical Analysis 1: Comparison: Group 1: Apremilast Immediate Release vs Group 1: Apremilast Modified Release 1; To compare each test formulation with the reference formulation in each group, an analysis of variance (ANOVA) was performed on the natural log-transformed Cmax value. The ANOVA model included treatment, sequence, and period as fixed effects and subject nested within sequence as a random effect; Test type: Other; Ratio of Adjusted Geometric Means = 65.3, 90% CI 2-sided [55.0 to 77.6] — Ratio of adjusted geometric means (Apremilast Modified Release 1 / Apremilast Immediate Release) expressed as a percentage
Statistical Analysis 2: Comparison: Group 1: Apremilast Immediate Release vs Group 1: Apremilast Modified Release 2; To compare each test formulation with the reference formulation in each group, an ANOVA was performed on the natural log-transformed Cmax value. The ANOVA model included treatment, sequence, and period as fixed effects and subject nested within sequence as a random effect; Test type: Other; Ratio of Adjusted Geometric Means = 80.4, 90% CI 2-sided [67.8 to 95.5] — Ratio of adjusted geometric means (Apremilast Modified Release 2 / Apremilast Immediate Release) expressed as a percentage
Statistical Analysis 3: Comparison: Group 1: Apremilast Immediate Release vs Group 1: Apremilast Modified Release 3; [analysis description as in outcome 1, analysis 2]; Test type: Other; Ratio of Adjusted Geometric Means = 84.2, 90% CI 2-sided [70.9 to 99.9] — Ratio of adjusted geometric means (Apremilast Modified Release 3 / Apremilast Immediate Release) expressed as a percentage

2. Secondary Outcome: Group 1: Number of Participants With Treatment-emergent Adverse Events
Description: An adverse event (AE) is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a participant during the course of a study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the participant's health, including laboratory test values, regardless of etiology.
  A treatment-emergent AE (TEAE) was defined as any AE that occurred after dosing of the study drug.
  A serious adverse event (SAE) is any AE occurring at any dose that:
  * Resulted in death;
  * Was life-threatening;
  * Required inpatient hospitalization or prolongation of existing hospitalization;
  * Resulted in persistent or significant disability/incapacity;
  * Was a congenital anomaly/birth defect;
  * Constituted an important medical event.
Time Frame: Adverse events were collected for 7 to 10 days after each treatment.
Population: Participants who received at least one dose of apremilast.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Apremilast Immediate Release | Group 1: Apremilast Modified Release 1 | Group 1: Apremilast Modified Release 2 | Group 1: Apremilast Modified Release 3
Number analyzed (Participants) | 16 | 16 | 16 | 16
Participants
  Any treatment-emergent adverse event (TEAE) | 5 | 4 | 2 | 1
  TEAEs related to study drug | 4 | 1 | 2 | 1
  Serious adverse events | 0 | 0 | 0 | 0
  Serious adverse events related to study drug | 0 | 0 | 0 | 0
  Discontinuations due to adverse events | 0 | 0 | 0 | 0
  Deaths | 0 | 0 | 0 | 0

3. Primary Outcome: Group 1: Area Under the Plasma Concentration-time Curve From Time Zero to the Last Measured Time Point (AUC0-t) of Apremilast
Description: as for outcome 1
Time Frame: as for outcome 1
Population: The PK population included all participants who received at least one dose of apremilast and had evaluable PK profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Group 1: Apremilast Immediate Release | Group 1: Apremilast Modified Release 1 | Group 1: Apremilast Modified Release 2 | Group 1: Apremilast Modified Release 3
Number analyzed (Participants) | 16 | 16 | 16 | 16
ng*h/mL | 6918.49 (47.7) | 4277.83 (88.2) | 4925.69 (67.7) | 5103.07 (54.3)
Statistical Analysis 1: Comparison: Group 1: Apremilast Immediate Release vs Group 1: Apremilast Modified Release 1; To compare each test formulation with the reference formulation in each group, an ANOVA was performed on the natural log-transformed AUC0-t value. The ANOVA model included treatment, sequence, and period as fixed effects and subject nested within sequence as a random effect; Test type: Other; Ratio of Adjusted Geometric Means = 61.8, 90% CI 2-sided [51.7 to 73.9] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Group 1: Apremilast Immediate Release vs Group 1: Apremilast Modified Release 2; [analysis description as in outcome 3, analysis 1]; Test type: Other; Ratio of Adjusted Geometric Means = 71.2, 90% CI 2-sided [59.6 to 85.1] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Group 1: Apremilast Immediate Release vs Group 1: Apremilast Modified Release 3; [analysis description as in outcome 3, analysis 1]; Test type: Other; Ratio of Adjusted Geometric Means = 73.8, 90% CI 2-sided [61.7 to 88.2] — [estimate comment as in outcome 1, analysis 3]

4. Primary Outcome: Group 1: Area Under the Plasma Concentration-time Curve From Time Zero Extrapolated to Infinity (AUC0-∞) of Apremilast
Description: as for outcome 1
Time Frame: as for outcome 1
Population: The PK population included all participants who received at least one dose of apremilast and had evaluable PK profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Group 1: Apremilast Immediate Release | Group 1: Apremilast Modified Release 1 | Group 1: Apremilast Modified Release 2 | Group 1: Apremilast Modified Release 3
Number analyzed (Participants) | 16 | 16 | 16 | 16
ng*h/mL | 6955.76 (47.9) | 4330.66 (88.2) | 4961.51 (67.8) | 5147.83 (54.5)
Statistical Analysis 1: Comparison: Group 1: Apremilast Immediate Release vs Group 1: Apremilast Modified Release 1; To compare each test formulation with the reference formulation in each group, an ANOVA was performed on the natural log-transformed AUC0-∞ value. The ANOVA model included treatment, sequence, and period as fixed effects and subject nested within sequence as a random effect; Test type: Other; Ratio of Adjusted Geometric Means = 62.3, 90% CI 2-sided [52.1 to 74.4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Group 1: Apremilast Immediate Release vs Group 1: Apremilast Modified Release 2; [analysis description as in outcome 4, analysis 1]; Test type: Other; Ratio of Adjusted Geometric Means = 71.3, 90% CI 2-sided [59.7 to 85.2] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Group 1: Apremilast Immediate Release vs Group 1: Apremilast Modified Release 3; [analysis description as in outcome 4, analysis 1]; Test type: Other; Ratio of Adjusted Geometric Means = 74.0, 90% CI 2-sided [62.0 to 88.4] — [estimate comment as in outcome 1, analysis 3]

5. Primary Outcome: Group 1: Time to Observed Maximum Plasma Concentration (Tmax) of Apremilast
Description: as for outcome 1
Time Frame: as for outcome 1
Population: The PK population included all participants who received at least one dose of apremilast and had evaluable PK profiles.
Measure: Median (Full Range); unit: hours
Arm/Group | Group 1: Apremilast Immediate Release | Group 1: Apremilast Modified Release 1 | Group 1: Apremilast Modified Release 2 | Group 1: Apremilast Modified Release 3
Number analyzed (Participants) | 16 | 16 | 16 | 16
hours | 3.00 [2.00 to 5.00] | 4.00 [2.00 to 8.00] | 4.00 [2.00 to 8.00] | 4.00 [3.00 to 14.00]
Statistical Analysis 1: Comparison: Group 1: Apremilast Immediate Release vs Group 1: Apremilast Modified Release 1; Tmax was analyzed by nonparametric methods. The median difference and 90% CI of the median difference were calculated from the Hodges-Lehrmann estimate; Test type: Other; p = 0.0090, Wilcoxon signed-rank test; Median Difference = 1.00, 90% CI 2-sided [0.5 to 2.00] — Median difference (Apremilast Modified Release 1 - Apremilast Immediate Release) calculated from the Hodges-Lehmann estimate
Statistical Analysis 2: Comparison: Group 1: Apremilast Immediate Release vs Group 1: Apremilast Modified Release 2; [analysis description as in outcome 5, analysis 1]; Test type: Other; p = 0.0073, Wilcoxon signed-rank test; Median Difference = 1.26, 90% CI 2-sided [0.50 to 3.00] — Median difference (Apremilast Modified Release 2 - Apremilast Immediate Release) calculated from the Hodges-Lehmann estimate
Statistical Analysis 3: Comparison: Group 1: Apremilast Immediate Release vs Group 1: Apremilast Modified Release 3; [analysis description as in outcome 5, analysis 1]; Test type: Other; p < 0.0001, Wilcoxon signed-rank test; Median Difference = 2.00, 90% CI 2-sided [1.00 to 3.00] — Median difference (Apremilast Modified Release 3 - Apremilast Immediate Release) calculated from the Hodges-Lehmann estimate

6. Primary Outcome: Group 1: Half-life of Apremilast in Terminal Phase (T1/2)
Description: as for outcome 1
Time Frame: as for outcome 1
Population: The PK population included all participants who received at least one dose of apremilast and had evaluable PK profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Group 1: Apremilast Immediate Release | Group 1: Apremilast Modified Release 1 | Group 1: Apremilast Modified Release 2 | Group 1: Apremilast Modified Release 3
Number analyzed (Participants) | 16 | 16 | 16 | 16
hours | 7.12 (23.3) | 7.43 (21.7) | 6.88 (22.0) | 7.29 (21.8)

7. Primary Outcome: Group 1: Apparent Total Plasma Clearance (CL/F) of Apremilast
Description: as for outcome 1
Time Frame: as for outcome 1
Population: The PK population included all participants who received at least one dose of apremilast and had evaluable PK profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Group 1: Apremilast Immediate Release | Group 1: Apremilast Modified Release 1 | Group 1: Apremilast Modified Release 2 | Group 1: Apremilast Modified Release 3
Number analyzed (Participants) | 16 | 16 | 16 | 16
L/h | 8.63 (47.9) | 17.32 (88.2) | 15.12 (67.8) | 14.57 (54.5)

8. Primary Outcome: Group 1: Apparent Total Volume of Distribution (Vz/F) of Apremilast
Description: as for outcome 1
Time Frame: as for outcome 1
Population: The PK population included all participants who received at least one dose of apremilast and had evaluable PK profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | Group 1: Apremilast Immediate Release | Group 1: Apremilast Modified Release 1 | Group 1: Apremilast Modified Release 2 | Group 1: Apremilast Modified Release 3
Number analyzed (Participants) | 16 | 16 | 16 | 16
liters | 88.65 (32.5) | 185.65 (64.7) | 149.97 (53.5) | 153.23 (34.8)

9. Primary Outcome: Group 1: Relative Bioavailability of Apremilast Test Formulations Relative to Reference Corrected by Dose
Description: Relative bioavailability of each test formulation compared to the reference formulation corrected by dose, calculated as:
  (AUC0-∞/Dose[test]) / (AUC0-∞/Dose[reference]) * 100%.
Time Frame: as for outcome 1
Population: The PK population included all participants who received at least one dose of apremilast and had evaluable PK profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percent availability
Arm/Group | Group 1: Apremilast Modified Release 1 | Group 1: Apremilast Modified Release 2 | Group 1: Apremilast Modified Release 3
Number analyzed (Participants) | 16 | 16 | 16
percent availability | 39.85 (53.7) | 45.65 (47.0) | 47.37 (22.9)

10. Primary Outcome: Group 1: Relative Bioavailability of Apremilast Test Formulations Relative to Reference
Description: Relative bioavailability of each test formulation compared to the reference formulation corrected by dose, calculated as:
  (AUC0-∞[test]) / (AUC0-∞[reference]) * 100%.
Time Frame: as for outcome 1
Population: The PK population included all participants who received at least one dose of apremilast and had evaluable PK profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percent availability
Arm/Group | Group 1: Apremilast Modified Release 1 | Group 1: Apremilast Modified Release 2 | Group 1: Apremilast Modified Release 3
Number analyzed (Participants) | 16 | 16 | 16
percent availability | 62.26 (53.7) | 71.33 (47.0) | 74.01 (22.9)

11. Primary Outcome: Group 2: Observed Maximum Plasma Concentration (Cmax) of Apremilast
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Group 2: Apremilast Immediate Release: Participants received two oral doses of 30 mg apremilast immediate release tablets 12 hours apart (reference formulation).
- Group 2: Apremilast Modified Release 4: Participants received a single oral dose 75 mg apremilast capsule prototype MR 4.
- Group 2: Apremilast Modified Release 5: Participants received a single oral dose 75 mg apremilast capsule prototype MR 5.
- Group 2: Apremilast Modified Release 6: Participants received a single oral dose 75 mg apremilast capsule prototype MR 6.
Arm/Group | Group 2: Apremilast Immediate Release | Group 2: Apremilast Modified Release 4 | Group 2: Apremilast Modified Release 5 | Group 2: Apremilast Modified Release 6
Number analyzed (Participants) | 16 | 16 | 16 | 16
ng/mL | 405.38 (30.2) | 368.45 (37.2) | 298.96 (34.1) | 325.20 (35.1)
Statistical Analysis 1: Comparison: Group 2: Apremilast Immediate Release vs Group 2: Apremilast Modified Release 4; [analysis description as in outcome 1, analysis 2]; Test type: Other; Ratio of Adjusted Geometric Means = 90.9, 90% CI 2-sided [81.8 to 101.1] — Ratio of adjusted geometric means (Apremilast Modified Release 4 / Apremilast Immediate Release) expressed as a percentage
Statistical Analysis 2: Comparison: Group 2: Apremilast Immediate Release vs Group 2: Apremilast Modified Release 5; [analysis description as in outcome 1, analysis 2]; Test type: Other; Ratio of Adjusted Geometric Means = 73.7, 90% CI 2-sided [66.3 to 82.0] — Ratio of adjusted geometric means (Apremilast Modified Release 5 / Apremilast Immediate Release) expressed as a percentage
Statistical Analysis 3: Comparison: Group 2: Apremilast Immediate Release vs Group 2: Apremilast Modified Release 6; [analysis description as in outcome 1, analysis 2]; Test type: Other; Ratio of Adjusted Geometric Means = 80.2, 90% CI 2-sided [72.2 to 89.2] — Ratio of adjusted geometric means (Apremilast Modified Release 6 / Apremilast Immediate Release) expressed as a percentage

12. Primary Outcome: Group 2: Area Under the Plasma Concentration-time Curve From Time Zero to the Last Measured Time Point (AUC0-t) of Apremilast
Description: as for outcome 1
Time Frame: as for outcome 1
Population: The PK population included all participants who received at least one dose of apremilast and had evaluable PK profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Group 2: Apremilast Immediate Release | Group 2: Apremilast Modified Release 4 | Group 2: Apremilast Modified Release 5 | Group 2: Apremilast Modified Release 6
Number analyzed (Participants) | 16 | 16 | 16 | 16
ng*h/mL | 6635.78 (35.9) | 5634.92 (40.2) | 4780.60 (39.3) | 5177.46 (36.9)
Statistical Analysis 1: Comparison: Group 2: Apremilast Immediate Release vs Group 2: Apremilast Modified Release 4; [analysis description as in outcome 3, analysis 1]; Test type: Other; Ratio of Adjusted Geometric Means = 84.9, 90% CI 2-sided [77.5 to 93.0] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 2: Comparison: Group 2: Apremilast Immediate Release vs Group 2: Apremilast Modified Release 5; [analysis description as in outcome 3, analysis 1]; Test type: Other; Ratio of Adjusted Geometric Means = 72.0, 90% CI 2-sided [65.8 to 78.9] — [estimate comment as in outcome 11, analysis 2]
Statistical Analysis 3: Comparison: Group 2: Apremilast Immediate Release vs Group 2: Apremilast Modified Release 6; [analysis description as in outcome 3, analysis 1]; Test type: Other; Ratio of Adjusted Geometric Means = 78.0, 90% CI 2-sided [71.2 to 85.5] — [estimate comment as in outcome 11, analysis 3]

13. Primary Outcome: Group 2: Area Under the Plasma Concentration-time Curve From Time Zero Extrapolated to Infinity (AUC0-∞) of Apremilast
Description: as for outcome 1
Time Frame: as for outcome 1
Population: The PK population included all participants who received at least one dose of apremilast and had evaluable PK profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Group 2: Apremilast Immediate Release | Group 2: Apremilast Modified Release 4 | Group 2: Apremilast Modified Release 5 | Group 2: Apremilast Modified Release 6
Number analyzed (Participants) | 16 | 16 | 16 | 16
ng*h/mL | 6669.26 (36.0) | 5700.66 (40.1) | 4843.46 (38.9) | 5259.40 (35.9)
Statistical Analysis 1: Comparison: Group 2: Apremilast Immediate Release vs Group 2: Apremilast Modified Release 4; [analysis description as in outcome 4, analysis 1]; Test type: Other; Ratio of Adjusted Geometric Means = 85.5, 90% CI 2-sided [78.1 to 93.6] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 2: Comparison: Group 2: Apremilast Immediate Release vs Group 2: Apremilast Modified Release 5; [analysis description as in outcome 4, analysis 1]; Test type: Other; Ratio of Adjusted Geometric Means = 72.6, 90% CI 2-sided [66.3 to 79.5] — [estimate comment as in outcome 11, analysis 2]
Statistical Analysis 3: Comparison: Group 2: Apremilast Immediate Release vs Group 2: Apremilast Modified Release 6; [analysis description as in outcome 4, analysis 1]; Test type: Other; Ratio of Adjusted Geometric Means = 78.9, 90% CI 2-sided [72.0 to 86.4] — [estimate comment as in outcome 11, analysis 3]

14. Primary Outcome: Group 2: Time to Observed Maximum Plasma Concentration (Tmax) of Apremilast
Description: as for outcome 1
Time Frame: as for outcome 1
Population: The PK population included all participants who received at least one dose of apremilast and had evaluable PK profiles.
Measure: Median (Full Range); unit: hours
Arm/Group | Group 2: Apremilast Immediate Release | Group 2: Apremilast Modified Release 4 | Group 2: Apremilast Modified Release 5 | Group 2: Apremilast Modified Release 6
Number analyzed (Participants) | 16 | 16 | 16 | 16
hours | 2.00 [1.00 to 3.00] | 4.00 [3.00 to 8.00] | 3.00 [2.00 to 6.00] | 4.00 [2.00 to 6.00]
Statistical Analysis 1: Comparison: Group 2: Apremilast Immediate Release vs Group 2: Apremilast Modified Release 4; [analysis description as in outcome 5, analysis 1]; Test type: Other; p = 0.0002, Wilcoxon signed-rank test; Median Difference = 2.00, 90% CI 2-sided [1.00 to 3.00] — Median difference (Apremilast Modified Release 4 - Apremilast Immediate Release) calculated from the Hodges-Lehmann estimate
Statistical Analysis 2: Comparison: Group 2: Apremilast Immediate Release vs Group 2: Apremilast Modified Release 5; [analysis description as in outcome 5, analysis 1]; Test type: Other; p = 0.0049, Wilcoxon signed-rank test; Median Difference = 1.02, 90% CI 2-sided [0.50 to 2.00] — Median difference (Apremilast Modified Release 5 - Apremilast Immediate Release) calculated from the Hodges-Lehmann estimate
Statistical Analysis 3: Comparison: Group 2: Apremilast Immediate Release vs Group 2: Apremilast Modified Release 6; [analysis description as in outcome 5, analysis 1]; Test type: Other; p = 0.0010, Wilcoxon signed-rank test; Median Difference = 1.50, 90% CI 2-sided [1.00 to 2.00] — Median difference (Apremilast Modified Release 6 - Apremilast Immediate Release) calculated from the Hodges-Lehmann estimate

15. Primary Outcome: Group 2: Half-life of Apremilast in Terminal Phase (T1/2)
Description: as for outcome 1
Time Frame: as for outcome 1
Population: The PK population included all participants who received at least one dose of apremilast and had evaluable PK profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Group 2: Apremilast Immediate Release | Group 2: Apremilast Modified Release 4 | Group 2: Apremilast Modified Release 5 | Group 2: Apremilast Modified Release 6
Number analyzed (Participants) | 16 | 16 | 16 | 16
hours | 8.16 (26.3) | 8.98 (22.9) | 8.43 (28.9) | 8.75 (29.6)

16. Primary Outcome: Group 2: Apparent Total Plasma Clearance (CL/F) of Apremilast
Description: as for outcome 1
Time Frame: as for outcome 1
Population: The PK population included all participants who received at least one dose of apremilast and had evaluable PK profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Group 2: Apremilast Immediate Release | Group 2: Apremilast Modified Release 4 | Group 2: Apremilast Modified Release 5 | Group 2: Apremilast Modified Release 6
Number analyzed (Participants) | 16 | 16 | 16 | 16
L/h | 9.00 (36.0) | 13.16 (40.1) | 15.48 (38.9) | 14.26 (35.9)

17. Primary Outcome: Group 2: Apparent Total Volume of Distribution (Vz/F) of Apremilast
Description: as for outcome 1
Time Frame: as for outcome 1
Population: The PK population included all participants who received at least one dose of apremilast and had evaluable PK profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | Group 2: Apremilast Immediate Release | Group 2: Apremilast Modified Release 4 | Group 2: Apremilast Modified Release 5 | Group 2: Apremilast Modified Release 6
Number analyzed (Participants) | 16 | 16 | 16 | 16
liters | 105.88 (35.3) | 170.51 (34.0) | 188.24 (37.5) | 180.10 (48.3)

18. Primary Outcome: Group 2: Relative Bioavailability of Apremilast Test Formulations Relative to Reference Corrected by Dose
Description: as for outcome 9
Time Frame: as for outcome 1
Population: The PK population included all participants who received at least one dose of apremilast and had evaluable PK profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percent availability
Arm/Group | Group 2: Apremilast Modified Release 4 | Group 2: Apremilast Modified Release 5 | Group 2: Apremilast Modified Release 6
Number analyzed (Participants) | 16 | 16 | 16
percent availability | 54.71 (26.0) | 46.48 (23.5) | 50.47 (13.2)

19. Primary Outcome: Group 2: Relative Bioavailability of Apremilast Test Formulations Relative to Reference
Description: as for outcome 10
Time Frame: as for outcome 1
Population: The PK population included all participants who received at least one dose of apremilast and had evaluable PK profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percent availability
Arm/Group | Group 2: Apremilast Modified Release 4 | Group 2: Apremilast Modified Release 5 | Group 2: Apremilast Modified Release 6
Number analyzed (Participants) | 16 | 16 | 16
percent availability | 85.48 (26.0) | 72.62 (23.5) | 78.86 (13.2)

20. Primary Outcome: Group 3: Observed Maximum Plasma Concentration (Cmax) of Apremilast
Description: as for outcome 1
Time Frame: as for outcome 1
Population: The PK population included all participants who received at least one dose of apremilast and had evaluable PK profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Group 3: Apremilast Immediate Release: Participants received two oral doses of 30 mg apremilast immediate release tablets 12 hours apart (reference formulation).
- Group 3: Apremilast Modified Release 8: Participants received a single oral dose 80 mg apremilast capsule prototype MR 8.
- Group 3: Apremilast Modified Release 9: Participants received a single oral dose 80 mg apremilast capsule prototype MR 9.
Arm/Group | Group 3: Apremilast Immediate Release | Group 3: Apremilast Modified Release 8 | Group 3: Apremilast Modified Release 9
Number analyzed (Participants) | 18 | 18 | 18
ng/mL | 378.59 (31.6) | 344.61 (28.7) | 334.51 (33.6)
Statistical Analysis 1: Comparison: Group 3: Apremilast Immediate Release vs Group 3: Apremilast Modified Release 8; [analysis description as in outcome 1, analysis 2]; Test type: Other; Ratio of Adjusted Geometric Means = 91.0, 90% CI 2-sided [80.4 to 103.0] — Ratio of adjusted geometric means (Apremilast Modified Release 8 / Apremilast Immediate Release) expressed as a percentage
Statistical Analysis 2: Comparison: Group 3: Apremilast Immediate Release vs Group 3: Apremilast Modified Release 9; [analysis description as in outcome 1, analysis 2]; Test type: Other; Ratio of Adjusted Geometric Means = 88.4, 90% CI 2-sided [78.1 to 100.0] — Ratio of adjusted geometric means (Apremilast Modified Release 9 / Apremilast Immediate Release) expressed as a percentage

21. Primary Outcome: Group 3: Area Under the Plasma Concentration-time Curve From Time Zero to the Last Measured Time Point (AUC0-t) of Apremilast
Description: as for outcome 1
Time Frame: as for outcome 1
Population: The PK population included all participants who received at least one dose of apremilast and had evaluable PK profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Group 3: Apremilast Immediate Release | Group 3: Apremilast Modified Release 8 | Group 3: Apremilast Modified Release 9
Number analyzed (Participants) | 18 | 18 | 18
ng*h/mL | 5493.38 (33.7) | 4427.56 (32.7) | 4310.62 (35.0)
Statistical Analysis 1: Comparison: Group 3: Apremilast Immediate Release vs Group 3: Apremilast Modified Release 8; [analysis description as in outcome 3, analysis 1]; Test type: Other; Ratio of Adjusted Geometric Means = 80.6, 90% CI 2-sided [73.8 to 88.0] — [estimate comment as in outcome 20, analysis 1]
Statistical Analysis 2: Comparison: Group 3: Apremilast Immediate Release vs Group 3: Apremilast Modified Release 9; [analysis description as in outcome 3, analysis 1]; Test type: Other; Ratio of Adjusted Geometric Means = 78.5, 90% CI 2-sided [71.9 to 85.7] — [estimate comment as in outcome 20, analysis 2]

22. Primary Outcome: Group 3: Area Under the Plasma Concentration-time Curve From Time Zero Extrapolated to Infinity (AUC0-∞) of Apremilast
Description: as for outcome 1
Time Frame: as for outcome 1
Population: The PK population included all participants who received at least one dose of apremilast and had evaluable PK profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Group 3: Apremilast Immediate Release | Group 3: Apremilast Modified Release 8 | Group 3: Apremilast Modified Release 9
Number analyzed (Participants) | 18 | 18 | 18
ng*h/mL | 5518.28 (33.8) | 4477.63 (32.7) | 4359.49 (35.0)
Statistical Analysis 1: Comparison: Group 3: Apremilast Immediate Release vs Group 3: Apremilast Modified Release 8; [analysis description as in outcome 4, analysis 1]; Test type: Other; Ratio of Adjusted Geometric Means = 81.1, 90% CI 2-sided [74.3 to 88.6] — [estimate comment as in outcome 20, analysis 1]
Statistical Analysis 2: Comparison: Group 3: Apremilast Immediate Release vs Group 3: Apremilast Modified Release 9; [analysis description as in outcome 4, analysis 1]; Test type: Other; Ratio of Adjusted Geometric Means = 79.0, 90% CI 2-sided [72.3 to 86.3] — [estimate comment as in outcome 20, analysis 2]

23. Primary Outcome: Group 3: Time to Observed Maximum Plasma Concentration (Tmax) of Apremilast
Description: as for outcome 1
Time Frame: as for outcome 1
Population: The PK population included all participants who received at least one dose of apremilast and had evaluable PK profiles.
Measure: Median (Full Range); unit: hours
Arm/Group | Group 3: Apremilast Immediate Release | Group 3: Apremilast Modified Release 8 | Group 3: Apremilast Modified Release 9
Number analyzed (Participants) | 18 | 18 | 18
hours | 3.00 [2.00 to 5.03] | 4.00 [2.00 to 6.00] | 4.00 [2.00 to 6.00]
Statistical Analysis 1: Comparison: Group 3: Apremilast Immediate Release vs Group 3: Apremilast Modified Release 8; [analysis description as in outcome 5, analysis 1]; Test type: Other; p = 0.0374, Wilcoxon signed-rank test; Median Difference = 0.98, 90% CI 2-sided [0.02 to 1.50] — Median difference (Apremilast Modified Release 8 - Apremilast Immediate Release) calculated from the Hodges-Lehmann estimate
Statistical Analysis 2: Comparison: Group 3: Apremilast Immediate Release vs Group 3: Apremilast Modified Release 9; [analysis description as in outcome 5, analysis 1]; Test type: Other; p = 0.1907, Wilcoxon signed-rank test; Median Difference = 0.51, 90% CI 2-sided [0.00 to 1.50] — Median difference (Apremilast Modified Release 9 - Apremilast Immediate Release) calculated from the Hodges-Lehmann estimate

24. Primary Outcome: Group 3: Half-life of Apremilast in Terminal Phase (T1/2)
Description: as for outcome 1
Time Frame: as for outcome 1
Population: The PK population included all participants who received at least one dose of apremilast and had evaluable PK profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Group 3: Apremilast Immediate Release | Group 3: Apremilast Modified Release 8 | Group 3: Apremilast Modified Release 9
Number analyzed (Participants) | 18 | 18 | 18
hours | 6.45 (23.8) | 6.58 (29.2) | 7.05 (27.0)

25. Primary Outcome: Group 3: Apparent Total Plasma Clearance (CL/F) of Apremilast
Description: as for outcome 1
Time Frame: as for outcome 1
Population: The PK population included all participants who received at least one dose of apremilast and had evaluable PK profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Group 3: Apremilast Immediate Release | Group 3: Apremilast Modified Release 8 | Group 3: Apremilast Modified Release 9
Number analyzed (Participants) | 18 | 18 | 18
L/h | 10.87 (33.8) | 17.87 (32.7) | 18.35 (35.0)

26. Primary Outcome: Group 2: Apparent Total Volume of Distribution (Vz/F) of Apremilast
Description: as for outcome 1
Time Frame: as for outcome 1
Population: The PK population included all participants who received at least one dose of apremilast and had evaluable PK profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | Group 3: Apremilast Immediate Release | Group 3: Apremilast Modified Release 8 | Group 3: Apremilast Modified Release 9
Number analyzed (Participants) | 18 | 18 | 18
liters | 101.23 (37.2) | 169.71 (34.0) | 186.69 (34.8)

27. Primary Outcome: Group 3: Relative Bioavailability of Apremilast Test Formulations Relative to Reference Corrected by Dose
Description: as for outcome 9
Time Frame: as for outcome 1
Population: The PK population included all participants who received at least one dose of apremilast and had evaluable PK profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percent availability
Arm/Group | Group 3: Apremilast Modified Release 8 | Group 3: Apremilast Modified Release 9
Number analyzed (Participants) | 18 | 18
percent availability | 45.64 (21.4) | 44.44 (21.1)

28. Primary Outcome: Group 3: Relative Bioavailability of Apremilast Test Formulations Relative to Reference
Description: as for outcome 10
Time Frame: as for outcome 1
Population: The PK population included all participants who received at least one dose of apremilast and had evaluable PK profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percent availability
Arm/Group | Group 3: Apremilast Modified Release 8 | Group 3: Apremilast Modified Release 9
Number analyzed (Participants) | 18 | 18
percent availability | 81.14 (21.4) | 79.00 (21.1)

29. Primary Outcome: Group 4: Observed Maximum Plasma Concentration (Cmax) of Apremilast
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Group 4: Apremilast Immediate Release: Participants received two oral doses of 30 mg apremilast immediate release tablets 12 hours apart (reference formulation).
- Group 4: Apremilast Modified Release 11: Participants received a single oral dose 80 mg apremilast capsule prototype MR 11.
- Group 4: Apremilast Modified Release 12: Participants received a single oral dose 80 mg apremilast capsule prototype MR 12.
- Group 4: Apremilast Modified Release 13: Participants received a single oral dose 80 mg apremilast capsule prototype MR 13.
- Group 4: Apremilast Modified Release 14: Participants received a single oral dose 80 mg apremilast capsule prototype MR 14.
Arm/Group | Group 4: Apremilast Immediate Release | Group 4: Apremilast Modified Release 11 | Group 4: Apremilast Modified Release 12 | Group 4: Apremilast Modified Release 13 | Group 4: Apremilast Modified Release 14
Number analyzed (Participants) | 29 | 29 | 28 | 28 | 28
ng/mL | 438.90 (29.1) | 480.59 (24.9) | 481.10 (29.3) | 316.43 (48.5) | 450.23 (32.5)
Statistical Analysis 1: Comparison: Group 4: Apremilast Immediate Release vs Group 4: Apremilast Modified Release 11; [analysis description as in outcome 1, analysis 2]; Test type: Other; Ratio of Adjusted Geometric Means = 109.4, 90% CI 2-sided [98.6 to 121.3] — Ratio of adjusted geometric means (Apremilast Modified Release 11 / Apremilast Immediate Release) expressed as a percentage
Statistical Analysis 2: Comparison: Group 4: Apremilast Immediate Release vs Group 4: Apremilast Modified Release 12; [analysis description as in outcome 1, analysis 2]; Test type: Other; Ratio of Adjusted Geometric Means = 107.2, 90% CI 2-sided [96.4 to 119.2] — Ratio of adjusted geometric means (Apremilast Modified Release 12 / Apremilast Immediate Release) expressed as a percentage
Statistical Analysis 3: Comparison: Group 4: Apremilast Immediate Release vs Group 4: Apremilast Modified Release 13; [analysis description as in outcome 1, analysis 2]; Test type: Other; Ratio of Adjusted Geometric Means = 72.7, 90% CI 2-sided [65.5 to 80.8] — Ratio of adjusted geometric means (Apremilast Modified Release 13 / Apremilast Immediate Release) expressed as a percentage
Statistical Analysis 4: Comparison: Group 4: Apremilast Immediate Release vs Group 4: Apremilast Modified Release 14; [analysis description as in outcome 1, analysis 2]; Test type: Other; Ratio of Adjusted Geometric Means = 103.5, 90% CI 2-sided [93.1 to 114.9] — Ratio of adjusted geometric means (Apremilast Modified Release 14 / Apremilast Immediate Release) expressed as a percentage

30. Primary Outcome: Group 4: Area Under the Plasma Concentration-time Curve From Time Zero to the Last Measured Time Point (AUC0-t) of Apremilast
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Group 4: Apremilast Immediate Release | Group 4: Apremilast Modified Release 11 | Group 4: Apremilast Modified Release 12 | Group 4: Apremilast Modified Release 13 | Group 4: Apremilast Modified Release 14
Number analyzed (Participants) | 29 | 29 | 28 | 28 | 28
ng*h/mL | 6976.02 (32.3) | 5701.21 (34.1) | 5811.24 (29.0) | 4700.70 (40.2) | 5324.80 (36.5)
Statistical Analysis 1: Comparison: Group 4: Apremilast Immediate Release vs Group 4: Apremilast Modified Release 11; [analysis description as in outcome 3, analysis 1]; Test type: Other; Ratio of Adjusted Geometric Means = 81.5, 90% CI 2-sided [75.2 to 88.3] — [estimate comment as in outcome 29, analysis 1]
Statistical Analysis 2: Comparison: Group 4: Apremilast Immediate Release vs Group 4: Apremilast Modified Release 12; [analysis description as in outcome 3, analysis 1]; Test type: Other; Ratio of Adjusted Geometric Means = 82.4, 90% CI 2-sided [75.9 to 89.5] — [estimate comment as in outcome 29, analysis 2]
Statistical Analysis 3: Comparison: Group 4: Apremilast Immediate Release vs Group 4: Apremilast Modified Release 13; [analysis description as in outcome 3, analysis 1]; Test type: Other; Ratio of Adjusted Geometric Means = 68.2, 90% CI 2-sided [62.9 to 74.0] — [estimate comment as in outcome 29, analysis 3]
Statistical Analysis 4: Comparison: Group 4: Apremilast Immediate Release vs Group 4: Apremilast Modified Release 14; [analysis description as in outcome 3, analysis 1]; Test type: Other; Ratio of Adjusted Geometric Means = 77.4, 90% CI 2-sided [71.3 to 84.0] — [estimate comment as in outcome 29, analysis 4]

31. Primary Outcome: Group 4: Area Under the Plasma Concentration-time Curve From Time Zero Extrapolated to Infinity (AUC0-∞) of Apremilast
Description: as for outcome 1
Time Frame: as for outcome 1
Population: The PK population included all participants who received at least one dose of apremilast and had evaluable PK profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Group 4: Apremilast Immediate Release | Group 4: Apremilast Modified Release 11 | Group 4: Apremilast Modified Release 12 | Group 4: Apremilast Modified Release 13 | Group 4: Apremilast Modified Release 14
Number analyzed (Participants) | 29 | 29 | 28 | 28 | 28
ng*h/mL | 7000.35 (32.2) | 5747.12 (34.0) | 5875.19 (28.6) | 4753.79 (40.1) | 5374.83 (36.8)
Statistical Analysis 1: Comparison: Group 4: Apremilast Immediate Release vs Group 4: Apremilast Modified Release 11; [analysis description as in outcome 4, analysis 1]; Test type: Other; Ratio of Adjusted Geometric Means = 81.9, 90% CI 2-sided [75.6 to 88.6] — [estimate comment as in outcome 29, analysis 1]
Statistical Analysis 2: Comparison: Group 4: Apremilast Immediate Release vs Group 4: Apremilast Modified Release 12; [analysis description as in outcome 4, analysis 1]; Test type: Other; Ratio of Adjusted Geometric Means = 83.0, 90% CI 2-sided [76.5 to 90.1] — [estimate comment as in outcome 29, analysis 2]
Statistical Analysis 3: Comparison: Group 4: Apremilast Immediate Release vs Group 4: Apremilast Modified Release 13; [analysis description as in outcome 4, analysis 1]; Test type: Other; Ratio of Adjusted Geometric Means = 68.8, 90% CI 2-sided [63.4 to 74.5] — [estimate comment as in outcome 29, analysis 3]
Statistical Analysis 4: Comparison: Group 4: Apremilast Immediate Release vs Group 4: Apremilast Modified Release 14; [analysis description as in outcome 4, analysis 1]; Test type: Other; Ratio of Adjusted Geometric Means = 77.8, 90% CI 2-sided [71.8 to 84.4] — [estimate comment as in outcome 29, analysis 4]

32. Primary Outcome: Group 4: Time to Observed Maximum Plasma Concentration (Tmax) of Apremilast
Description: as for outcome 1
Time Frame: as for outcome 1
Population: The PK population included all participants who received at least one dose of apremilast and had evaluable PK profiles.
Measure: Median (Full Range); unit: hours
Arm/Group | Group 4: Apremilast Immediate Release | Group 4: Apremilast Modified Release 11 | Group 4: Apremilast Modified Release 12 | Group 4: Apremilast Modified Release 13 | Group 4: Apremilast Modified Release 14
Number analyzed (Participants) | 29 | 29 | 28 | 28 | 28
hours | 3.00 [1.00 to 5.08] | 4.00 [2.00 to 6.00] | 4.00 [2.00 to 6.00] | 4.01 [2.00 to 14.00] | 3.52 [2.00 to 6.00]
Statistical Analysis 1: Comparison: Group 4: Apremilast Immediate Release vs Group 4: Apremilast Modified Release 11; [analysis description as in outcome 5, analysis 1]; Test type: Other; p = 0.0523, Wilcoxon signed-rank test; Median Difference = 0.98, 90% CI 2-sided [0.03 to 1.50] — Median difference (Apremilast Modified Release 11 - Apremilast Immediate Release) calculated from the Hodges-Lehmann estimate
Statistical Analysis 2: Comparison: Group 4: Apremilast Immediate Release vs Group 4: Apremilast Modified Release 12; [analysis description as in outcome 5, analysis 1]; Test type: Other; p = 0.2598, Wilcoxon signed-rank test; Median Difference = 0.50, 90% CI 2-sided [0.00 to 1.00] — Median difference (Apremilast Modified Release 12 - Apremilast Immediate Release) calculated from the Hodges-Lehmann estimate
Statistical Analysis 3: Comparison: Group 4: Apremilast Immediate Release vs Group 4: Apremilast Modified Release 13; [analysis description as in outcome 5, analysis 1]; Test type: Other; p = 0.0053, Wilcoxon signed-rank test; Median Difference = 1.50, 90% CI 2-sided [1.00 to 3.00] — Median difference (Apremilast Modified Release 13 - Apremilast Immediate Release) calculated from the Hodges-Lehmann estimate
Statistical Analysis 4: Comparison: Group 4: Apremilast Immediate Release vs Group 4: Apremilast Modified Release 14; [analysis description as in outcome 5, analysis 1]; Test type: Other; p = 0.1093, Wilcoxon signed-rank test; Median Difference = 0.50, 90% CI 2-sided [0.00 to 1.00] — Median difference (Apremilast Modified Release 14 - Apremilast Immediate Release) calculated from the Hodges-Lehmann estimate

33. Primary Outcome: Group 4: Half-life of Apremilast in Terminal Phase (T1/2)
Description: as for outcome 1
Time Frame: as for outcome 1
Population: The PK population included all participants who received at least one dose of apremilast and had evaluable PK profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Group 4: Apremilast Immediate Release | Group 4: Apremilast Modified Release 11 | Group 4: Apremilast Modified Release 12 | Group 4: Apremilast Modified Release 13 | Group 4: Apremilast Modified Release 14
Number analyzed (Participants) | 29 | 29 | 28 | 28 | 28
hours | 6.25 (24.8) | 7.40 (25.2) | 7.51 (34.9) | 7.09 (31.0) | 7.13 (32.5)

34. Primary Outcome: Group 4: Apparent Total Plasma Clearance (CL/F) of Apremilast
Description: as for outcome 1
Time Frame: as for outcome 1
Population: The PK population included all participants who received at least one dose of apremilast and had evaluable PK profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Group 4: Apremilast Immediate Release | Group 4: Apremilast Modified Release 11 | Group 4: Apremilast Modified Release 12 | Group 4: Apremilast Modified Release 13 | Group 4: Apremilast Modified Release 14
Number analyzed (Participants) | 29 | 29 | 28 | 28 | 28
L/h | 8.57 (32.2) | 13.92 (34.0) | 13.62 (28.6) | 16.83 (40.1) | 14.88 (36.8)

35. Primary Outcome: Group 4: Apparent Total Volume of Distribution (Vz/F) of Apremilast
Description: as for outcome 1
Time Frame: as for outcome 1
Population: The PK population included all participants who received at least one dose of apremilast and had evaluable PK profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | Group 4: Apremilast Immediate Release | Group 4: Apremilast Modified Release 11 | Group 4: Apremilast Modified Release 12 | Group 4: Apremilast Modified Release 13 | Group 4: Apremilast Modified Release 14
Number analyzed (Participants) | 29 | 29 | 28 | 28 | 28
liters | 77.30 (36.0) | 148.66 (32.5) | 147.59 (41.5) | 172.16 (44.6) | 153.18 (36.1)

36. Primary Outcome: Group 4: Relative Bioavailability of Apremilast Test Formulations Relative to Reference Corrected by Dose
Description: as for outcome 9
Time Frame: as for outcome 1
Population: The PK population included all participants who received at least one dose of apremilast and had evaluable PK profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percent availability
Arm/Group | Group 4: Apremilast Modified Release 11 | Group 4: Apremilast Modified Release 12 | Group 4: Apremilast Modified Release 13 | Group 4: Apremilast Modified Release 14
Number analyzed (Participants) | 29 | 27 | 28 | 28
percent availability | 46.18 (22.3) | 46.86 (27.7) | 38.65 (34.0) | 43.70 (26.9)

37. Primary Outcome: Group 4: Relative Bioavailability of Apremilast Test Formulations Relative to Reference
Description: as for outcome 10
Time Frame: as for outcome 1
Population: The PK population included all participants who received at least one dose of apremilast and had evaluable PK profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percent availability
Arm/Group | Group 4: Apremilast Modified Release 11 | Group 4: Apremilast Modified Release 12 | Group 4: Apremilast Modified Release 13 | Group 4: Apremilast Modified Release 14
Number analyzed (Participants) | 29 | 27 | 28 | 28
percent availability | 82.10 (22.3) | 83.31 (27.7) | 68.71 (34.0) | 77.68 (26.9)

38. Secondary Outcome: Group 2: Number of Participants With Treatment-emergent Adverse Events
Description: as for outcome 2
Time Frame: Adverse events were collected for 7 to 10 days after each treatment.
Population: Participants who received at least one dose of apremilast.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 2: Apremilast Immediate Release | Group 2: Apremilast Modified Release 4 | Group 2: Apremilast Modified Release 5 | Group 2: Apremilast Modified Release 6
Number analyzed (Participants) | 16 | 16 | 16 | 16
Participants
  Any treatment-emergent adverse event (TEAE) | 4 | 4 | 6 | 5
  TEAEs related to study drug | 4 | 2 | 5 | 4
  Serious adverse events | 0 | 0 | 0 | 0
  Serious adverse events related to study drug | 0 | 0 | 0 | 0
  Discontinuations due to adverse events | 0 | 0 | 0 | 0
  Deaths | 0 | 0 | 0 | 0

39. Secondary Outcome: Group 3: Number of Participants With Treatment-emergent Adverse Events
Description: as for outcome 2
Time Frame: Adverse events were collected for 7 to 10 days after each treatment.
Population: Participants who received at least one dose of apremilast.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 3: Apremilast Immediate Release | Group 3: Apremilast Modified Release 8 | Group 3: Apremilast Modified Release 9
Number analyzed (Participants) | 18 | 18 | 18
Participants
  Any treatment-emergent adverse event (TEAE) | 5 | 3 | 3
  TEAEs related to study drug | 1 | 0 | 2
  Serious adverse events | 0 | 0 | 0
  Serious adverse events related to study drug | 0 | 0 | 0
  Discontinuations due to adverse events | 0 | 0 | 0
  Deaths | 0 | 0 | 0

40. Secondary Outcome: Group 4: Number of Participants With Treatment-emergent Adverse Events
Description: as for outcome 2
Time Frame: Adverse events were collected for 7 to 10 days after each treatment.
Population: Participants who received at least one dose of apremilast.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 4: Apremilast Immediate Release | Group 4: Apremilast Modified Release 11 | Group 4: Apremilast Modified Release 12 | Group 4: Apremilast Modified Release 13 | Group 4: Apremilast Modified Release 14
Number analyzed (Participants) | 29 | 29 | 28 | 28 | 28
Participants
  Any treatment-emergent adverse event (TEAE) | 13 | 7 | 7 | 7 | 9
  TEAE related to study drug | 9 | 7 | 6 | 6 | 7
  Serious adverse events | 0 | 0 | 0 | 0 | 0
  Serious adverse events related to study drug | 0 | 0 | 0 | 0 | 0
  Discontinuation due to adverse events | 0 | 0 | 0 | 0 | 0
  Deaths | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected for 7 to 10 days after each treatment.
Description: Adverse events are reported for all participants who received at least one dose of apremilast.
Groups:
- Group 1 Total: Participants received the following 4 treatments, given in 4 possible sequences (ADBC, BACD, CBDA, and DCAB) with 7 to 10 days between each treatment:
  A) Two oral doses of 30 mg apremilast immediate release tablets 12 hours apart (reference formulation) B) A single oral dose 75 mg apremilast tablet prototype MR 1 C) A single oral dose 75 mg apremilast tablet prototype MR 2 D) A single oral dose 75 mg apremilast capsule prototype MR 3.
- Group 2 Total: Participants received the following 4 treatments, given in 4 possible sequences (AGEF, EAFG, FEGA, and GFAE) with 7 to 10 days between each treatment:
  A) Two oral doses of 30 mg apremilast immediate release tablets 12 hours apart (reference formulation) E) A single oral dose 75 mg apremilast capsule prototype MR 4 F) A single oral dose 75 mg apremilast capsule prototype MR 5 G) A single oral dose 75 mg apremilast capsule prototype MR 6
- Group 3 Total: Participants received the following 3 treatments, given in 6 possible sequences (AIJ, IJA, JAI, AJI, IAJ, or JIA) with 7 to 10 days between each treatment:
  A) Two oral doses of 30 mg apremilast immediate release tablets 12 hours apart (reference formulation) I) A single oral dose 80 mg apremilast capsule prototype MR 8 J) A single oral dose 80 mg apremilast capsule prototype MR 9
- Group 4 Total: Participants received the following 5 treatments, given in 10 possible sequences (ALOMN, LMANO, MNLOA, NOMAL, OANLM, NMOLA, ONAML, AOLNM, LAMON, or MLNAO) with 7 to 10 days between each treatment:
  A) Two oral doses of 30 mg apremilast immediate release tablets 12 hours apart (reference formulation) L) A single oral dose 80 mg apremilast capsule prototype MR 11 M) A single oral dose 80 mg apremilast capsule prototype MR 12 N) A single oral dose 80 mg apremilast capsule prototype MR 13 O) A single oral dose 80 mg apremilast capsule prototype MR 14
- Overall Total: All participants who received any dose of apremilast during the study.
Arm/Group | Group 1: Apremilast Immediate Release | Group 1: Apremilast Modified Release 1 | Group 1: Apremilast Modified Release 2 | Group 1: Apremilast Modified Release 3 | Group 1 Total | Group 2: Apremilast Immediate Release | Group 2: Apremilast Modified Release 4 | Group 2: Apremilast Modified Release 5 | Group 2: Apremilast Modified Release 6 | Group 2 Total | Group 3: Apremilast Immediate Release | Group 3: Apremilast Modified Release 8 | Group 3: Apremilast Modified Release 9 | Group 3 Total | Group 4: Apremilast Immediate Release | Group 4: Apremilast Modified Release 11 | Group 4: Apremilast Modified Release 12 | Group 4: Apremilast Modified Release 13 | Group 4: Apremilast Modified Release 14 | Group 4 Total | Overall Total
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/16 | 0/16 | 0/16 | 0/16 | 0/16 | 0/16 | 0/16 | 0/18 | 0/18 | 0/18 | 0/18 | 0/29 | 0/29 | 0/28 | 0/28 | 0/28 | 0/30 | 0/80
Other Adverse Events (participants affected / at risk) | 5/16 | 4/16 | 2/16 | 1/16 | 8/16 | 4/16 | 4/16 | 6/16 | 5/16 | 8/16 | 5/18 | 3/18 | 3/18 | 7/18 | 12/29 | 5/29 | 7/28 | 5/28 | 7/28 | 17/30 | 40/80
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: Apremilast Immediate Release (N=16) | Group 1: Apremilast Modified Release 1 (N=16) | Group 1: Apremilast Modified Release 2 (N=16) | Group 1: Apremilast Modified Release 3 (N=16) | Group 1 Total (N=16) | Group 2: Apremilast Immediate Release (N=16) | Group 2: Apremilast Modified Release 4 (N=16) | Group 2: Apremilast Modified Release 5 (N=16) | Group 2: Apremilast Modified Release 6 (N=16) | Group 2 Total (N=16) | Group 3: Apremilast Immediate Release (N=18) | Group 3: Apremilast Modified Release 8 (N=18) | Group 3: Apremilast Modified Release 9 (N=18) | Group 3 Total (N=18) | Group 4: Apremilast Immediate Release (N=29) | Group 4: Apremilast Modified Release 11 (N=29) | Group 4: Apremilast Modified Release 12 (N=28) | Group 4: Apremilast Modified Release 13 (N=28) | Group 4: Apremilast Modified Release 14 (N=28) | Group 4 Total (N=30) | Overall Total (N=80)
CONJUNCTIVAL HYPERAEMIA (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
VISION BLURRED (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 2 | 5 | 7
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 2
CHANGE OF BOWEL HABIT (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
DIARRHOEA (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 3 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 3 | 6
DRY MOUTH (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
HAEMORRHOIDS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
NAUSEA (Gastrointestinal disorders) | 2 | 0 | 1 | 1 | 2 | 0 | 0 | 3 | 1 | 3 | 1 | 0 | 1 | 2 | 1 | 2 | 1 | 0 | 0 | 4 | 11
FOLLICULITIS (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
GASTROENTERITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 3
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 3 | 3
ARTHROPOD STING (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
LACERATION (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 3
PROCEDURAL COMPLICATION (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 2
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 2 | 3
PROCEDURAL SITE REACTION (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 3 | 1 | 0 | 0 | 0 | 0 | 1 | 5
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2
DIZZINESS (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 2 | 2 | 4 | 5 | 6
DYSGEUSIA (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
HEADACHE (Nervous system disorders) | 3 | 1 | 2 | 0 | 4 | 3 | 0 | 2 | 1 | 5 | 0 | 0 | 0 | 0 | 8 | 4 | 4 | 3 | 4 | 13 | 22
PRESYNCOPE (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 3
SYNCOPE (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
DRY THROAT (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
ERYTHEMA (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.